CLINICAL TRIAL: NCT06520878
Title: Impact of NANO-PSO (omega 5) Supplementation on Cognitive Abilities of Older Adults with Mild to Moderate Non-vascular Cognitive Impairment
Brief Title: Impact of NANO-PSO on Cognition in Older Adults with Mild to Moderate Cognitive Impairment
Acronym: COGMEG5
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Distribuidora Biolife SA de CV (Industry)
Responsible Party: Principal Investigator, Alejandro Padilla Isassi, Principal researcher of the geriatrics area, Distribuidora Biolife SA de CV
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENS-2024-TL001
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cognition
Keywords: NANO-PSO; Omega 5; Supplementation; Cognitive impairment; Antioxidants
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Nano-PSO

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NANO-PSO (Experimental): 640 mg of NANO-PSO (pomegranate seed oil)
  Interventions: Dietary Supplement: NANO-PSO (pomegranate seed oil)
- Mineral oil (Placebo Comparator): 640 mg of mineral oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NANO-PSO (pomegranate seed oil) — NANO-PSO administered orally, 2 capsules, equivalent to 640 mg of pomegranate seed oil, every 24 hours in the morning with food.
  Other Names: Granagard; Omega 5
  Arms: NANO-PSO
Dietary Supplement: Placebo — Placebo administered orally, 2 capsules, equivalent to 640 mg of mineral oil, every 24 hours in the morning with food.
  Arms: Mineral oil

SUMMARY:
The objective of this randomized, triple-blind, placebo-controlled clinical trial is to compare NANO-PSO therapy against placebo in improving cognitive abilities in older adults with mild to moderate non-vascular cognitive impairment over six months of treatment. The primary questions it aims to answer are:

• Does NANO-PSO therapy improve cognitive abilities in older adults with mild to moderate non-vascular cognitive impairment over six months of treatment compared to placebo?

The researchers will compare NANO-PSO therapy against placebo to see if it benefits the cognitive abilities of geriatric patients.

Participants will be required to:

* Consume two capsules of NANO-PSO or placebo daily in the morning for six months.
* Be evaluated monthly by phone to identify potential risks and ensure adherence to the treatment.
* Be evaluated in person at 90 and 180 days of treatment.
* The patient or primary caregiver must maintain a log to confirm daily dose consumption and will have a direct communication line with the attending physicians in case of questions about ingestion or possible adverse reactions.
* At the end of the final patient evaluation, a quality questionnaire will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients attended at the Hospital Español.
* Patients of any gender who are 60 years or older.
* Patients presenting with mild to moderate cognitive impairment.
* Meet the diagnostic criteria for "probable dementia" of the National Institute on Aging and the Alzheimer's Association (NIA-AA) (2011).
* Meet the criteria for the typical variant of Alzheimer's disease, specifically a specific clinical phenotype.
* Progressive and gradual change in memory functions reported by the patient or the informant for at least 6 months.
* Objective evidence of a hippocampal-type amnesic syndrome, based on significant impairment in the performance of episodic memory tests with established specificity for AD.
* Subjects are primary and secondary school graduates and have the ability to complete cognitive capacity tests and other specified tests in the program.
* Total score on the Hachinski Ischemic Scale (HIS) ≤ 4.
* Patients who sign the informed consent.

Exclusion Criteria:

* Patients with known allergy to any component of the NANO-PSO capsule (e.g., fish).
* Patients with short bowel syndrome, bariatric surgery, or gluten reaction that may affect intestinal absorption.
* Patients in palliative care with a life expectancy of less than 6 months according to the NECPAL scale.
* Patients with terminality criteria established in the comprehensive palliative care management guide of Mexico.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive status assessment | Assessed at baseline, 3, and 6 months.
  Cognitive status assessment using the Mini-Mental State Examination, which ranges from 0 to 30 points and the higher score is better with higher cognition

SECONDARY OUTCOMES:
Patients' fatigue status | Assessed at baseline, 3, and 6 months.
  Evaluation using the 9-item Fatigue Severity Scale, which measures the severity of fatigue and its impact on the daily activities and lifestyle of patients. The scale ranges from 9 to 63 points and the higher the score, the worse the feeling of fatigue
Selective attention and processing speed | Assessed at baseline, 3, and 6 months.
  Selective attention and processing speed will be evaluated using the Trail Making Test (TMT), where the average time for TMT Part A is 29 seconds, with more than 78 seconds being considered deficient. For TMT Part B, the average time is 75 seconds, and more than 273 seconds is considered deficient.
Frailty | Assessed at baseline, 3, and 6 months.
  Frailty will be assessed using the Fried Frailty Criteria (Phenotype Model), which comprises five criteria. Based on these criteria. 0 criteria = No frailty; 1 to 2 criteria = Pre-frailty; 3 or more criteria = Frailty

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Padilla Isassi, Geriatrician and researcher, Principal Investigator — Distribuidora Biolife S.A. de C.V.
Locations (1):
- Hospital Español. Av Ejercito Nacional 613, Miguel Hidalgo, CDMX, 11520, Miguel Hidalgo, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Sharing the information has not been considered or thought of due to the confidentiality statuses of the Hospital Español

REFERENCES:
- [Background] Binyamin O, Nitzan K, Frid K, Ungar Y, Rosenmann H, Gabizon R. Brain targeting of 9c,11t-Conjugated Linoleic Acid, a natural calpain inhibitor, preserves memory and reduces Abeta and P25 accumulation in 5XFAD mice. Sci Rep. 2019 Dec 5;9(1):18437. doi: 10.1038/s41598-019-54971-9. PMID 31804596